CLINICAL TRIAL: NCT05216198
Title: Evaluation of the Effectiveness of a City Hospital Care Network for the Care of Patients With Transient Ischemic Accident (TIA)
Acronym: AIT-AMBU-GRE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: EssaiClinique_AIT-AMBU-GRE
Record Dates: First submitted 2022-01-11; First posted 2022-01-31 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-01

CONDITIONS: Transient Ischemic Attack
Keywords: transient ischemic attack; neurovascular unit; managed care program
MeSH Terms: conditions — Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TIA patients: Diagnostic of TIA by the exams performed in the emergencies of CHUGA.
  Interventions: Other: Check of the different exams performed at the emergencies

INTERVENTIONS:
Other: Check of the different exams performed at the emergencies — Check of the different exams performed at the emergencies

SUMMARY:
Transient ischemic accidents (TIA) are a frequent resort to hospitalization in the emergency department and are serious events in terms of recurrence and handicap. The organization of the "TIA sector" at CHUGA aims to facilitate on the one hand the care of the patient during his hospitalization in the emergencies and on the other hand to allow a safer discharge of the patient as well as his follow-up in ambulatory. The aim of this study is to study the feasibility of comprehensive short-term outpatient management after hospitalization in the emergencies. The research hypothesis is that 90% of patients complete all of the 10 recommended examinations for the diagnosis of TIA, analysis of its risk factors and initiation of necessary treatments, if necessary.

DETAILED DESCRIPTION:
Current knowledge on pathology Transient ischemic accidents (TIA) are a frequent resort to hospitalization in the emergency department (378 visits in 2019 to the CHUGA emergencies, 340 in 2020, or about 1 entry for this reason per day) and are serious events in terms of recurrence and handicap. The risk of Cerebral Vascular Accident (stroke) is around 10% at 3 months after the first episode of TIA [1]. Standardizing care and improving patient compliance with treatment and monitoring of their pathology aims to reduce the recurrence and the occurrence of more serious consequences.

In 2021, the Northern Alpine Emergency Network (RENAU) published standardized care for all hospitals and clinics dependent on this network, based on the French recommendations of the Haute Autorité de Santé and the French Neurovascular Society (SFNV).

This care was put in place at the Emergency Department of the CHU Grenoble Alpes (CHUGA) in the form of an "TIA program" and defines the patient's journey when he presents signs compatible with the suspicion of TIA. In addition to being based on national and regional recommendations, this sector has been improved by providing a questionnaire to all Neuro-Vascular Units (NVU) in France.

The organization of the "TIA sector" at CHUGA aims to facilitate on the one hand the care of the patient during his hospitalization in the emergency room and on the other hand to allow a safer discharge of the patient as well as his follow-up in ambulatory.

For example, a Parisian study, carried out at the Bichat hospital [2], showed that a standardized treatment pathway for TIAs was linked to a reduction of more than 30% in the risk of stroke 3 months after the TIA.

On arrival at the Emergency Department, in the event of any suggestive signs, the patient is included in the "TIA sector". He is examined as quickly as possible by an emergency physician and / or the neurologist on call. A predefined biology is taken and an electrocardiogram (ECG) is performed.

The patient undergoes a brain imaging test. Depending on availability, two imaging modalities are possible: brain CT-scan without injection followed by Doppler ultrasound of the supra-aortic trunks during the week during working hours, or a CT angiography with visualization of the supra-aortic trunks at night, on weekends and on holidays. Finally, the patient benefits from close monitoring. Depending on the clinical evaluation and the examinations carried out, the neurologist based in the Emergency Department, in agreement with the emergency physician, decides on the continuation of the treatment (hospitalization / come back home, drug treatment).

The criteria for hospitalization are generally represented by the discovery of a cardiac arrhythmia, an abnormality in the brain imaging or supra-aortic trunks, repeated TIAs, a significant duration of symptoms or a history and important cardiovascular risk factors.

If the patient does not present criteria for hospitalization, a return home is offered. For 56% of patients at the CHUGA in 2019 and 62% in 2020, outpatient care was decided. These are the patients that interest us in this study. When discharging from the emergency room, the "outpatient" treatment route is relatively heavy. Treatment will eventually be initiated and the patient will have outpatient examinations as well as schedule several consultations.

The patient must in particular schedule a consultation with a cardiologist (to perform a Holter ECG and a cardiac ultrasound), carry out several additional examinations including a brain MRI and laboratory tests and schedule a follow-up with a neurologist and his attending physician. .

The aim of this study is to study the feasibility of comprehensive short-term outpatient management after hospitalization in the emergencies. We want to assess the proper performance of all the examinations prescribed from the Emergency Department, the taking of the prescribed treatment, the patient's understanding of his pathology and his feelings about his care.

Patient management is not affected by this study.

Depending on the results, we will be able to target if certain elements are not feasible and thus improve the sector or even distribute it to other centers, in particular via the RENAU.

It is a single-center prospective descriptive epidemiological study conducted at the CHUGA within the Emergency Department.

Research hypotheses and expected results The research hypothesis is that 90% of patients complete all of the 10 recommended examinations for the diagnosis of TIA, analysis of its risk factors and initiation of necessary treatments, if necessary.

This percentage is arbitrary because no such study on the subject has yet been published. This high rate seems relevant to us to reflect the proper functioning of the sector.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization in the Emergency Department of the CHUGA for suspicion of TIA
* Possible or probable TIA diagnosis on discharge
* Major patient
* Outpatient care after emergency care

Exclusion Criteria:

* Protected patient (guardianship, curatorship, people not affiliated with Social Security)
* Patient deprived of liberty by a judicial or administrative decision
* Patient hospitalized without consent under Articles L. 3212-1 and L. 3213-1 which does not fall under the provisions of Article L. 1121-8
* Adult patient subject to a legal protection measure or unable to express consent
* Pregnant, lactating or parturient women
* Patient who does not speak French
* Inability to answer the phone to answer questions
* No attending physician

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Diagnostic of TIA by the exams performed in the emergencies of CHUGA.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
The objective of the research is to study the feasibility of outpatient treatment for TIA from the emergency room, by evaluating the percentage of patients who have completed 100% of the additional examinations included in the course. | 6 months
  The primary endpoint is the mandatory completion of the 10 items recommended by the SFNV and the RENAU, as part of the diagnosis and management of TIA:
  1. Recommended standard biology (including assessment of cardiovascular risk factors)
  2. The electrocardiogram
  3. Brain imaging
  4. Imaging of the supraortic trunks
  5. The summary of all examinations by a neurologist
  6. The introduction of antiplatelet therapy
  7. The introduction of statins
  8. The follow-up consultation with the attending physician in the month following discharge from the emergency room.
  9. Consultation with a cardiologist, with performance of an echocardiography and a Holter ECG
  10. Performing a brain MRI

SECONDARY OUTCOMES:
Identify the additional examinations that are not performed during the patient's care, and the difficulties in carrying out the standardized care offered to the Emergency Department | 6 months
  Collection of examinations not performed during patient care
Evaluate the patient's adherence and understanding to the care sector | 6 months
  Assessment of the patient's adherence to and understanding of the sector, based on a score on 8 questions rated from 0 to 5 Use of the score in questions V of the questionnaire to assess the patient's feelings
Identify the barriers to membership in the care sector | 6 months
  Collection and interpretation of examinations not performed during patient care
Identify complications at one month including a recurrence of TIA or stroke | 6 months
  Occurrence of a complication at one month (TIA or stroke) on the declarative basis, by the patient, during the telephone call one month after discharge from the Emergency Department

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble Alpes - Urgences, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Amarenco P, Benavente O. EXPRESS transient ischemic attack study: speed the process! Stroke. 2008 Aug;39(8):2400-1. doi: 10.1161/STROKEAHA.108.514166. Epub 2008 Jul 3. No abstract available. PMID 18599804
- [Background] Amarenco P. Not all patients should be admitted to the hospital for observation after a transient ischemic attack. Stroke. 2012 May;43(5):1448-9. doi: 10.1161/STROKEAHA.111.636753. No abstract available. PMID 22529312
- [Background] Amarenco P, Lavallee PC, Monteiro Tavares L, Labreuche J, Albers GW, Abboud H, Anticoli S, Audebert H, Bornstein NM, Caplan LR, Correia M, Donnan GA, Ferro JM, Gongora-Rivera F, Heide W, Hennerici MG, Kelly PJ, Kral M, Lin HF, Molina C, Park JM, Purroy F, Rothwell PM, Segura T, Skoloudik D, Steg PG, Touboul PJ, Uchiyama S, Vicaut E, Wang Y, Wong LKS; TIAregistry.org Investigators. Five-Year Risk of Stroke after TIA or Minor Ischemic Stroke. N Engl J Med. 2018 Jun 7;378(23):2182-2190. doi: 10.1056/NEJMoa1802712. Epub 2018 May 16. PMID 29766771
- [Background] Lavallee PC, Meseguer E, Abboud H, Cabrejo L, Olivot JM, Simon O, Mazighi M, Nifle C, Niclot P, Lapergue B, Klein IF, Brochet E, Steg PG, Leseche G, Labreuche J, Touboul PJ, Amarenco P. A transient ischaemic attack clinic with round-the-clock access (SOS-TIA): feasibility and effects. Lancet Neurol. 2007 Nov;6(11):953-60. doi: 10.1016/S1474-4422(07)70248-X. PMID 17928270
- [Background] Cucchiara BL, Kasner SE. All patients should be admitted to the hospital after a transient ischemic attack. Stroke. 2012 May;43(5):1446-7. doi: 10.1161/STROKEAHA.111.636746. No abstract available. PMID 22529311